CLINICAL TRIAL: NCT06099561
Title: Svårbehandlat självskadebeteende-Vilka Insatser är Effektiva?
Brief Title: Intractable Self-harm-What Support is Effective?
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: Department of Psychology. Lund University. (Unknown); Department of Clinical Sciences, Malmö. Faculty of Medicine, Lund University. (Unknown)
Responsible Party: Sponsor
Other Study IDs: Dnr 2023-01650-01
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Self-harm
Keywords: Deliberate self-harm; Suicide
MeSH Terms: conditions — Self-Injurious Behavior; Suicide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Individuals with current severe, imminent and lethal self-harm with a history of at least two interventions without sufficient reduction of self-harm or suffering.
  Interventions: Behavioral: National specialized medical care unit for severe self-harm behaviour-Consultation model

INTERVENTIONS:
Behavioral: National specialized medical care unit for severe self-harm behaviour-Consultation model — Extensive assessments. Consultation and training for existing treatment providers and caregivers. Network-meetings for providers and caregivers.

SUMMARY:
The aim of this project is to evaluate a novel treatment program for individuals with intractable and lethal self-harm.

The main questions are:

1: Is there, in individuals with intractable self-harm, a relevant improvement in daily functioning and is this improvement related to the provided interventions?

The secondary research questions are:

2. Is there, in individuals with intractable self-harm, a relevant improvement in frequency and severity of self-harm?

3. Is there, in individuals with intractable self-harm, a relevant improvement in voluntary hospital admissions?

4. Is there, in individuals with intractable self-harm, a relevant improvement in compulsary hospital admissions?

5. Is there, in individuals with intractable self-harm, a relevant improvement in the use of medication pro re nata?

6. Is there, in individuals with intractable self-harm, a relevant improvement in cost-effectiveness related to the provided interventions?

DETAILED DESCRIPTION:
Individuals with intractable, imminent and lethal self-harm often have multifaceted psychiatric symptoms, pervasive suffering, high mortality and a reduced level of daily functioning. Severe self-harm can lead to long periods of psychiatric inpatient care which can lead to reduced autonomy and aggravated self-harm. Effects of this care remain uncertain. The Swedish National Board of Welfare has provided National specialized medical care units for severe self-harm behaviour to three Swedish hospitals.

In one of this hospitals, Region Skåne, the intervention will be consultation-based. Individuals with intractable self-harm will be offered an assessment and review of all medical records which will result in a individualized intervention plan. Interventions include further assessments and supporting the existing treatment providers, families or caregivers. Recurring network-meetings will occur every three months as well as at he end of the intervention.

Data collection will include self-report measures as well as information from charts and national och regional registries.

ELIGIBILITY:
Inclusion Criteria:

* Having tried or made serious attempt to try at least two different interventions with evidence to reduce self-harm, without sufficient reduction in suffering or self-harm

Exclusion Criteria:

* Need for translation services to complete measures or interviews
* Not able to complete measures or interviews

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A group of individuals with severe self-harm, commonly with comorbid psychiatric diagnoses and cognitive challanges.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The World Health Organization Disability Assessment Schedule II (WHODAS 2.0) | Monthly from baseline to endpointat 24 months and at follow-up at 36 months.
  Level of daily functioning and disability in the domains of cognition, mobility, self-care, getting along with other people and life activities.

SECONDARY OUTCOMES:
Five Self-harm behaviour groupings measure (5S-HM) | Weekly from baseline to endpointat 24 months and at follow-up at 36 months.
  Indirect and direct self-harming behaviour
The 5-level EQ-5D | Monthly from baseline to endpointat 24 months and at follow-up at 36 months.
  Quality of life scale
Cost effectiveness | Monthly from baseline to endpointat 24 months and at follow-up at 36 months.
  Quantities and costs related to healthcare, municipal, social and rescue services.

CONTACTS AND LOCATIONS:
Locations (1):
- National Highly Specialized Unit for Self-Harm Behaviours, Skåne, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Possible ot applicable due to Swedish data protection legislation.